CLINICAL TRIAL: NCT04435769
Title: Non-interventional Study Describing Direct Costs Related to Anticoagulation Treatment in Patients With Nonvalvular Atrial Fibrillation (NVAF) in Secondary Stroke Prevention Prescribed Apixaban or Warfarin Treatment
Brief Title: Non-Interventional Study Describing Direct Costs Related to Anti-coagulation Treatment
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B0661121; APIXABAN SECOND LINE (Other: Alias Study Number)
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-valvular Atrial Fibrillation (NVAF) on warfarin: The study follows two cohorts of Non-valvular Atrial Fibrillation (NVAF) patients, who used warfarin as a secondary stroke/TIA prevention.
- Non-valvular Atrial Fibrillation (NVAF) on apixaban: The study follows two cohorts of Non-valvular Atrial Fibrillation (NVAF) patients, who used apixaban as a secondary stroke/TIA prevention.

SUMMARY:
To describe the direct costs related to warfarin/apixaban treatment

DETAILED DESCRIPTION:
To describe the direct costs related to warfarin/apixaban treatment during the first 6 months of the secondary stroke prevention in NVAF patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-valvular atrial fibrillation (NVAF);
* New initiation of anticoagulation therapy (apixaban or warfarin) due to the ischemic event (stroke/TIA) meaning patients previously not anticoagulated due to diagnosis of NVAF;
* Indication to anticoagulation therapy as a secondary stroke prevention within 7 to 30 days after the stroke/TIA event;
* Apixaban arm: genetically determined higher sensitivity to warfarin;
* Patients whose status allowed oral treatment with apixaban/warfarin;
* Age ≥ 18;
* Access to patient´s records of the first 6 months of the warfarin/apixaban treatment.

Exclusion Criteria:

* Diagnosis of valvular disease;
* Treatment with other anticoagulants in previous 6 months due to other the NVAF indication;
* Treatment or prophylaxis of deep vein thrombosis or pulmonary embolism;
* Contraindications according SmPC of Eliquis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NVAF patients, who used either warfarin or apixaban as a secondary stroke/TIA prevention.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Fakultní nemocnice Motol, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B0661121

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data from eligible participants with non-valvular atrial fibrillation (NVAF) who started treatment with warfarin or apixaban for the prevention of a secondary stroke or transient ischemic attack (TIA) between 2009 to 2019 were observed in this study. Participants' records were retrieved and observed only for first 6 months of the warfarin/apixaban treatment. Collected data from all the participants were observed approximately for 10 months in this observational study.
Groups:
- Apixaban: Participants with NVAF who received apixaban as per clinical practice in real world for the prevention of a secondary stroke or TIA were observed during this retrospective study.
- Warfarin: Participants with NVAF who received warfarin as per clinical practice in real world for the prevention of a secondary stroke or TIA were observed during this retrospective study.
Period: Overall Study
Arm/Group | Apixaban | Warfarin
Started | 42 | 67
Full Analysis Set (FAS) | 42 | 67
Per Protocol (PP) Population | 40 | 63
Completed | 42 | 67
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: PP population comprised of participants who followed visit 2 schedule at 6 months (+/- 10 weeks), met all inclusion criteria and did not meet any of the exclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Apixaban | Warfarin | Total
Number analyzed (Participants) | 40 | 63 | 103
Age, Continuous [Mean (Standard Deviation); unit: Years] | 78.1 (12.1) | 79.5 (9.3) | 79.0 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 34 | 51
  Male | 23 | 29 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body-Mass Index (BMI) [Mean (Standard Deviation); unit: Kilogram per meter square (kg/m^2)] | 26.9 (4.8) | 28.7 (5.4) | 28.0 (5.2)
Duration from index event to the initiation of non-vitamin K antagonist anticoagulant therapy (NOAC) [Mean (Standard Deviation); unit: Days] — The index event was the first stroke/TIA event based on which the NOAC treatment was initiated.
  Days | 11.8 (12.7) | 10.0 (6.2) | 10.7 (9.2)
Number of Participants With Anticoagulant Treatment Before the Initiation of NOAC Therapy [Count of Participants; unit: Participants]
  Aspirin | 19 | 35 | 54
  Clopidogrel | 11 | 8 | 19
  Thrombolytics | 15 | 9 | 24
  Clexane | 18 | 26 | 44
  Fraxiparine | 14 | 19 | 33
  Low molecular weight heparin (LMWH) - preventive dose | 18 | 33 | 51

OUTCOME MEASURES:

1. Primary Outcome: CHA2-DS2-VASc Score at Baseline
Description: CHA2DS2-VASc scoring scale was used to estimate the risk of stroke and systemic emboli in participants with NVAF. CHA2DS2-VASc score was calculated based on 8 risk factors (age 65-74 years, age >=75 years, sex category, i.e. female sex, congestive heart failure history, hypertension history, stroke/TIA/thromboembolism history, vascular disease history and diabetes mellitus history). Total CHA2DS2-VASc score ranged from 0-9 where 0= low risk and 9= high risk of stroke.
Time Frame: Baseline (from retrospective data retrieved in the study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 40 | 63
Units on a scale | 4.6 (1.5) | 4.3 (1.7)

2. Primary Outcome: HAS-BLED Score at Baseline
Description: HAS-BLED scoring scale was used to estimate the risk of bleeding. HAS-BLED score was calculated based on 9 risk factors (hypertension, renal disease, liver disease, stroke history, prior major bleeding or predisposition to bleeding, labile international normalized ratio (INR), age >65 years, medication usage predisposing to bleeding and alcohol use). Total HAS-BLED score ranged from 0 to 9 where 0 = low risk and >=3 = high risk of bleed.
Time Frame: Baseline (from retrospective data retrieved in the study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 40 | 63
Units on a scale | 2.7 (1.2) | 2.5 (1.1)

3. Primary Outcome: CHA2-DS2-VASc Score at Month 6
Description: CHA2DS2-VASc scoring scale was used to estimate the risk of stroke and systemic emboli in participants with NVAF. CHA2DS2-VASc score was calculated based on 8 risk factors (age 65-74 years, age >=75 years, sex category i.e. female sex, congestive heart failure history, hypertension history, stroke/TIA/thromboembolism history, vascular disease history and diabetes mellitus history). Total CHA2DS2-VASc score ranged from 0-9 where 0= low risk and 9= high risk of stroke.
Time Frame: Month 6 (from retrospective data retrieved in the study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 40 | 63
Units on a scale | 5.0 (1.4) | 4.9 (1.4)

4. Primary Outcome: HAS-BLED Score at Month 6
Description: as for outcome 2
Time Frame: Month 6 (from retrospective data retrieved in the study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 40 | 63
Units on a scale | 3.1 (1.1) | 2.8 (1.3)

5. Primary Outcome: Percentage of Participants Categorized According to Number of Outpatient Visits During First 6 Months of Treatment
Description: In this outcome measure, percentage of participants were categorized according to number of outpatient visits from 0 to 5.
Time Frame: Up to first 6 months of treatment (from retrospective data retrieved in the study)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 40 | 63
Percentage of participants
  0 visit | 55.0 | 44.4
  1 visit | 32.5 | 36.5
  2 visits | 12.5 | 9.5
  3 visits | 0.0 | 3.2
  4 visits | 0.0 | 4.8
  5 visits | 0.0 | 1.6

6. Primary Outcome: Cost of Outpatient Visits During First 6 Months of Treatment
Description: Costs of outpatient visits were calculated for the first 6 months of treatment as the number of visits multiplied by the cost of the visit (450.0 Czech koruna [CZK] per visit). Costs were calculated based on the number of outpatient visits during the treatment.
Time Frame: Up to first 6 months of treatment (from retrospective data retrieved in the study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Czech koruna
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 40 | 63
Czech koruna | 258.8 (320.4) | 414.3 (525.7)

7. Primary Outcome: Percentage of Participants Categorized According to Number of International Normalized Ratios (INR) Measurements During First 6 Months of Treatment
Description: INR was defined as the ratio of the participant's prothrombin time and the normal mean prothrombin time. Prothrombin time defined as a time taken by the blood to clot in participants receiving oral anticoagulant medication. In this outcome measure, percentage of participants were categorized according to number of INR measurements included zero (0), 1 to 9, 10 to 19 and greater than or equal to (>=) 20.
Time Frame: Up to first 6 months of treatment (from retrospective data retrieved in the study)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 40 | 63
Percentage of participants
  0 | 97.5 | 0.0
  1 to 9 | 2.5 | 4.8
  10 to 19 | 0.0 | 46.0
  >=20 | 0.0 | 49.2

8. Primary Outcome: Cost of INR Measurements During First 6 Months of Treatment
Description: INR was defined as the ratio of the participant's prothrombin time and the normal mean prothrombin time. Prothrombin time defined as a time taken by the blood to clot in participants receiving oral anticoagulant medication. Costs related to INR measurements, were calculated for the period of 6 months as the number of INR measurements multiplied by the cost of the INR measurement (213.0 CZK per measurement). Costs were based on the expenditure of total number of INR measurements during first 6-month treatment.
Time Frame: Up to first 6 months of treatment (from retrospective data retrieved in the study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Czech koruna
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 40 | 63
Czech koruna | 5.3 (33.7) | 4003.0 (1230.2)

9. Primary Outcome: Dosage of Warfarin and Apixaban at the Initiation of the Treatment
Description: In this outcome measure, dosage of apixaban and warfarin used at the initiation of treatment was reported.
Time Frame: Baseline (from retrospective data retrieved in the study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Milligrams per day
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 40 | 63
Milligrams per day | 7.5 (2.5) | 5.9 (3.2)

10. Primary Outcome: Dosage of Warfarin and Apixaban During First 6 Months of Treatment
Description: In this outcome measure, dosage of apixaban and warfarin used during first 6 months of treatment was reported.
Time Frame: Up to first 6 months of treatment (from retrospective data retrieved in the study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Milligrams per day
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 40 | 63
Milligrams per day | 7.4 (2.5) | 4.6 (1.8)

11. Primary Outcome: Cost of Medication During First 6 Months of Treatment
Description: In this outcome measure, cost of medication, i.e., costs of apixaban and warfarin were based on the dosage of active substance and were calculated for the first 6 months of treatment (daily cost times 182.4 days), regardless of how long the individual participant treated was reported.
Time Frame: Up to first 6 months of treatment (from retrospective data retrieved in the study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Czech koruna
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 40 | 63
Czech koruna | 8551.0 (2932.5) | 1263.5 (0.0)

12. Primary Outcome: Percentage of Participants Categorized According to Number of Hospital Admissions
Description: In this outcome measure, percentage of participants were categorized according to number of hospital admissions from 0 to 3 were reported.
Time Frame: Up to first 6 months of treatment (from retrospective data retrieved in the study)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 40 | 63
Percentage of participants
  0 | 95.0 | 81.0
  1 | 2.5 | 14.3
  2 | 0.0 | 4.8
  3 | 2.5 | 0.0

13. Primary Outcome: Cost of Hospital Admissions During First 6 Months of Treatment
Description: In this outcome measure, costs of hospital admissions were based on the number of hospital admissions during the treatment period by considering the reason for hospitalization. If the reason for admission was not related to the recorded event (ischemic, hemorrhagic, or other adverse event), or the participant experienced none of these events, the cost of hospitalization was calculated as the number of days multiplied by the cost per a day of hospitalization (1898.2 CZK per day).
Time Frame: Up to first 6 months of treatment (from retrospective data retrieved in the study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Czech koruna
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 40 | 63
Czech koruna | 2777.5 (13820.1) | 12326.8 (43596.2)

14. Primary Outcome: Percentage of Participants Categorized According to Number of Diagnostic Procedures
Description: In this outcome measure, percentage of participants were categorized according to number of diagnostic procedures.
Time Frame: Up to first 6 months of treatment (from retrospective data retrieved in the study)
Population: Data collected by trial sites for diagnostic procedures were incorrect, hence data was not evaluated and analyzed for this outcome measure.
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 0 | 0

15. Primary Outcome: Percentage of Participants Categorized According to Type of Ischemic Events During First 6 Months of Treatment
Description: In this outcome measure, percentage of participants were categorized according to type of ischemic events which included cardiac ischemia and stroke/TIA.
Time Frame: Up to first 6 months of treatment (from retrospective data retrieved in the study)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 40 | 63
Percentage of participants
  Cardiac ischemia | 2.5 | 0.0
  Stroke/TIA | 0.0 | 9.5

16. Primary Outcome: Cost of Ischemic Events During First 6 Months of Treatment
Description: Costs of ischemic events (cardiac ischemia and stroke/TIA) included expenditure of diagnosis, medication, outpatient visits and hospitalization were reported based on the recorded number of ischemic events during the first 6 months of treatment.
Time Frame: Up to first 6 months of treatment (from retrospective data retrieved in the study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Czech koruna
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 40 | 63
Czech koruna | 684.8 (4331.2) | 5386.6 (16735.9)

17. Primary Outcome: Percentage of Participants Categorized With Major Hemorrhagic Events During First 6 Months of Treatment
Description: In this outcome measure, percentage of participants with major hemorrhagic events which included intracranial bleeding was reported.
Time Frame: Up to first 6 months of treatment (from retrospective data retrieved in the study)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 40 | 63
Percentage of participants | 2.5 | 3.2

18. Primary Outcome: Percentage of Participants Categorized According to Type of Minor Hemorrhagic Events During First 6 Months of Treatment
Description: In this outcome measure, percentage of participants were categorized according to type of minor hemorrhagic events which included epistaxis, gastrointestinal (GI) bleeding, muscle hematomas and intraparenchymal hematoma of the lower lobe.
Time Frame: Up to first 6 months of treatment (from retrospective data retrieved in the study)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 40 | 63
Percentage of participants
  Epistaxis | 2.5 | 0.0
  GI bleeding | 0.0 | 1.6
  Muscle hematomas | 2.5 | 0.0
  Other- Intraparenchymal hematoma of the lower lobe | 0.0 | 1.6

19. Primary Outcome: Cost of Major Hemorrhagic Events During First 6 Months of Treatment
Description: Costs of major hemorrhagic events (intracranial bleeding) included expenditure of diagnosis, medication, outpatient visits and hospitalization were reported based on the recorded number of major hemorrhagic events during the first 6 months of treatment.
Time Frame: Up to first 6 months of treatment (from retrospective data retrieved in the study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Czech koruna
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 40 | 63
Czech koruna | 2092.7 (13235.4) | 2657.4 (14793.8)

20. Primary Outcome: Cost of Minor Hemorrhagic Events During First 6 Months of Treatment
Description: Costs of minor hemorrhagic events (epistaxis, GI bleeding, muscle hematomas and intraparenchymal hematoma of the lower lobe) included expenditure of diagnosis, medication, outpatient visits and hospitalization were reported based on the recorded number of minor hemorrhagic events during the first 6 months of treatment.
Time Frame: Up to first 6 months of treatment (from retrospective data retrieved in the study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Czech koruna
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 40 | 63
Czech koruna | 1285.1 (5697.5) | 1666.7 (10157.1)

21. Primary Outcome: Number of Participants With Other Adverse Events During First 6 Months of Treatment
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Other adverse events included all events other than ischemic, major and minor hemorrhagic events.
Time Frame: Up to first 6 months of treatment (from retrospective data retrieved in the study)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 40 | 63
Participants | 2 | 1

22. Primary Outcome: Cost of Other Adverse Events During First 6 Months of Treatment
Description: Costs of other adverse events included expenditure of diagnosis, medication, outpatient visits and hospitalization were reported based on the number of other adverse events during the treatment.
Time Frame: Up to first 6 months of treatment (from retrospective data retrieved in the study)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Czech koruna
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 40 | 63
Czech koruna | 2063.9 (9628.8) | 1328.7 (10546.2)

23. Primary Outcome: Percentage of Participants Who Died (Treatment-Related) During First 6 Months of Treatment
Description: In this outcome measure, percentage of participants who died due to the given treatment were reported.
Time Frame: Up to first 6 months of treatment (from retrospective data retrieved in the study)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 40 | 63
Percentage of participants | 0.0 | 1.6

ADVERSE EVENTS:
Time Frame: 6 Months (from retrospective data retrieved in the study)
Description: An AE term may be reported as both a serious and non-serious AE, but are distinct events. An AE may be serious for 1 participant and non-serious for another participant, or a participant may have experienced both a serious and non-serious episode of the same event. FAS population defined as records from all participants collected into the study were included. Events were recorded from participants' clinical practice hospital documents. No medical dictionary was utilized in this study.
Arm/Group | Apixaban | Warfarin
All-Cause Mortality (participants affected / at risk) | 0/42 | 1/67
Serious Adverse Events (participants affected / at risk) | 2/42 | 10/67
Other Adverse Events (participants affected / at risk) | 4/42 | 0/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban (N=42) | Warfarin (N=67)
Cardiac ischemia (General disorders) | 1 | 0
Stroke/TIA (General disorders) | 0 | 6
Intracranial bleeding (General disorders) | 1 | 2
GI bleeding (General disorders) | 0 | 1
Intraparenchymal hematoma of the lower lobe (General disorders) | 0 | 1
Diarrhoea (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban (N=42) | Warfarin (N=67)
Epistaxis (General disorders) | 1 | 0
Muscle hematomas (General disorders) | 1 | 0
Feeling sick (General disorders) | 1 | 0
Headache (General disorders) | 1 | 0
Vertigo (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT04435769/Prot_SAP_000.pdf